CLINICAL TRIAL: NCT04805307
Title: An Open-Label, Phase 1, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of CMG901 in Subjects With Advanced Unresectable or Metastatic Solid Tumor
Brief Title: Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy, Phase 1 Study of CMG901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KYM901
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor; Gastric Cancer(Including Gastroesophageal Junction Adenocarcinoma); Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Part A：Dose Escalation: Modified 3+3 dose escalation design: an accelerated dose titration design followed by traditional 3+3 dose escalation design.
  Part B：Dose Expansion: Subjects will be enrolled at 2.2 mg/kg, 2.6 mg/kg, 3.0 mg/kg and/or other higher dose levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A, Dose escalation (Experimental): CMG901 will be administered in treatment cycles once every 3 weeks (Q3W). Dose escalation will be carried out according to a modified 3+3 dose-escalation design. Accelerated dose titration design will be used for the first 2 dose levels (0.3mg/kg and 0.6mg/kg), and then traditional 3+3 dose escalation design will be used for the following levels (1.2mg/kg, 1.8mg/kg, 2.2mg/kg, 2.6mg/kg and 3.0mg/kg).
  Interventions: Drug: CMG901
- Part B, Dose expansion,2.2mg/kg (Experimental): This cohort will comprise subjects with Claudin 18.2 positive gastric cancer (including gastroesophageal junction adenocarcinoma), pancreatic cancer, and other solid cancer with prior failure of, progression on, or intolerance to, standard therapy.
  Interventions: Drug: CMG901
- art B, Dose expansion,3.0mg/kg (Experimental): This cohort will comprise subjects with Claudin 18.2 positive gastric cancer (including gastroesophageal junction adenocarcinoma), pancreatic cancer, and other solid cancer with prior failure of, progression on, or intolerance to, standard therapy.
  Interventions: Drug: CMG901
- Part B, Dose expansion,3.0mg/kg (Experimental): This cohort will comprise subjects with Claudin 18.2 positive gastric cancer (including gastroesophageal junction adenocarcinoma), pancreatic cancer, and other solid cancer with prior failure of, progression on, or intolerance to, standard therapy.
  Interventions: Drug: CMG901

INTERVENTIONS:
Drug: CMG901 — CMG901 will be administered intravenously (IV) on Day 1 of every 21-day cycle. Individual subjects may continue study treatment until confirmed Progressive Disease(PD), unacceptable toxicity, initiation of new anti-tumor therapy, withdrawal from the study, or death, whichever occurs first.

SUMMARY:
This is a multi-center, open-label, dose escalation and dose expansion, Phase 1 study to evaluate the safety, tolerability, PK and preliminary anti-tumor activity of CMG901.

The dose escalation phase (Part A) will determine the MTD of CMG901 in subjects with relapsed and/or refractory advanced solid tumor for which there is no available standard therapy likely to confer clinical benefit, or the subject is not a candidate for such available therapy based on a modified 3+3 dose escalation design (an accelerated dose titration design followed by traditional 3+3 dose escalation design).

The dose expansion phase (Part B) will be conducted in subjects with advanced solid cancer with failure of standard treatment or no standard treatment who are Claudin 18.2 positive to preliminarily explore the efficacy and to determine the RP2D of CMG901.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with histologically or cytologically confirmed advanced solid tumors, who have failed to respond to standard of care (progression after treatment or intolerance) or who have no available standard of care regimen.
* Part A: Must provide archival tumor tissue specimen or agree to undergo a fresh biopsy if archival specimen is unavailable for retrospective Claudin 18.2 testing prior to enrollment;Subjects enrolled in Part A are not required to be positive for Claudin 18.2.
* Part A: Measurable or evaluable lesions per RECIST v 1.1.Part B: At least one measurable lesion per RECIST v1.1.
* Part B: Subjects shall provide fresh or archival tumor tissue samples before enrollment for assessment of Claudin 18.2 expression level (central laboratory) and should be positive for Claudin 18.2 as determined by the central laboratory. If the subject can provide positive Claudin 18.2 expression results which had been reported by the same central laboratory using the same method, there is no need for another test.
* Women of childbearing potential and male subjects must agree to remain abstinent or use contraceptive methods as defined by the protocol.
* Eastern Cooperative Oncology Group Performance Status 0-1.
* Side effects of any prior therapy or procedures for any medical condition has recovered to NCI-CTCAE v.5.0 Grade ≤ 1 or stable status by investigator.

Key Exclusion Criteria:

* Received: chemotherapy or any investigational anti-tumor agents within 28 days of the start of CMG901 treatment; molecularly-targeted agents, immunoconjugate, or antibody drug conjugate within 28 days or or 5 half-lives (whichever is shorter) of the start of CMG901 treatment; major surgery within 28 days of the start of CMG901 treatment; radiotherapy within 21 days of the start of CMG901 treatment; potent cytochrome P450 3A4 (CYP3A4) inhibitors within 14 days or or 5 half-lives (whichever is longer) of the start of CMG901 treatment.
* Diagnosis of immunodeficiency or requiring another form of chronic immunosuppressive therapy. Or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone or equivalent) within 7 days prior to the first dose.
* History of severe hypersensitivity to any component or excipient of CMG901.
* Ongoing or active infection or interstitial pneumonia assessed by investigator.
* Any severe cardiac dysfunction including left ventricular ejection fraction <50%, congestive heart failure ≥Grade 2 (New York Heart Association), QTc >480 msec, major cardiovascular and cerebrovascular diseases (e.g., congestive cardiac failure, acute myocardial infarction, unstable angina, stroke, transient ischemic attack, deep vein thrombosis or pulmonary embolism) within 6 months prior to the first dose of study drug.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Subjects with uncontrolled ascites, pleural effusion, or pericardial effusion by investigator.
* Preexisting sensory and/or motor neuropathy Grade ≥2.
* Uncontrolled diabetes mellitus or diabetic neuropathy within 3 months of the first dose of CMG901.
* Subjects with active hepatitis B or C, i.e., positive for anti-HCV antibody and positive for HCV RNA, or positive for HBsAg with detectable positive for HBV DNA (i.e., ≥ 2000 IU/mL).
* Any other conditions such as medical history, treatment, laboratory abnormalities that may confound the study results, interfere with the subject's compliance, or impair the interests of the subject, as assessed by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence of adverse events.Abnormal laboratory parameters, vital signs, 12-lead electrocardiogram and physical examination. Occurrence of Dose-limiting toxicity | Up to 30 days post the last dose, initiation of new anti-tumor therapy, withdrawal from the study, or death, whichever occurs first. DLTs are up to 21 days after the first dose
Part A: To determine the maximum tolerated dose (MTD) of CMG901 | Up to 21 days after the first dose
Part B: To preliminarily evaluate the Objective Response Rate (ORR) per RECIST v1.1 of CMG901 in subjects with Claudin 18.2-positive advanced solid cancer | Up to 24 months
Part B: Recommended phase II dose | Up to 24 months

SECONDARY OUTCOMES:
Part A & Part B: Area Under the Curve from 0 to the time of the last measurable concentration [AUC(0-last)] | 21 days after the first dose
Part A & Part B: Area Under the Curve over a dosing interval [AUC(0-tau)] | 21 days after the first dose
Part A & Part B: Area Under the Curve from 0 to infinity [AUC(0-inf)] | 21 days after the first dose
Part A & Part B: Peak Plasma Concentration (Cmax) | 21 days after the first dose
Part A & Part B: Time of Maximum Observed Concentration (Tmax) | 21 days after the first dose
Part A & Part B: Terminal elimination half-life (t1/2) | 21 days after the first dose
Part A & Part B: Clearance (CL) | 21 days after the first dose
Part A & Part B: Volume of distribution (Vz) | 21 days after the first dose
Part A & Part B: Observed concentration at the end of a dosing interval(Ctrough) | 21 days after the first dose
Part A & Part B: Area Under the Curve from 0 to the time of the last measurable concentration [AUC(0-last)] | up to 24 months
Part A & Part B: Area Under the Curve over a dosing interval [AUC(0-tau)] | up to 24 months
Part A & Part B: Peak Plasma Concentration (Cmax) | up to 24 months
Time of maximum observed concentration (Tmax) | up to 24 months
Part A & Part B: Terminal elimination half-life (t1/2) | up to 24 months
Part A & Part B: Clearance (CL) | up to 24 months
Part A & Part B: Volume of distribution (Vz) | up to 24 months
Part A & Part B: Volume of distribution at steady-state (Vss) | up to 24 months
Part A & Part B: Minimum concentration (Cmin) | up to 24 months
Part A & Part B: Observed concentration at the end of a dosing interval (Ctrough) | up to 24 months
Part A & Part B: Accumulation ratios of peak plasma concentration (Cmax) for multiple doses | up to 24 months
Part A & Part B: Accumulation ratios of area under the curve over a dosing interval [AUC(0-tau)] for multiple doses | up to 24 months
Part A & Part B: Incidence of anti-CMG901 | up to 24 months
Part A & Part B: Disease Control Rate (DCR) per RECIST v1.1 | up to 24 months
Part A & Part B: Duration of Response (DoR) per RECIST v1.1 | up to 24 months
Part A & Part B: Progression Free Survival (PFS) per RECIST v1.1 | up to 24 months
Part A&B:To evaluate the correlation between clinical efficacy of CMG901 and Claudin 18.2 expression | up to 24 months
Part A: Objective Response Rate (ORR) per RECIST v1.1 | up to 24 months
Part A & Part B: Overall Survival (OS) | up to 24 months
Part B: Incidence of adverse events graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Abnormal laboratory parameters, vital signs, 12-lead electrocardiogram and physical examination | Up to 30 days post the last dose, initiation of new anti-tumor therapy, withdrawal from the study, or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Sun Yat-sen University
Locations (32):
- China (32):
  - Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Hebei University, Baoding
  - Hunan Cancer Hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Cancer Hosppital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The Second Hospital of Anhui Medical University, Hefei
  - Affiliated Hospital of Jining Medical University, Jining
  - Lanzhou University Second Hospital, Lanzhou
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang
  - Meizhou People's Hospital, Meizhou
  - Jiangxi Cancer Hospital, Nanchang
  - Huashan Hospital, Fudan University, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - The Forth Hospital of Hebei Medical University and Hebei Tumor Hospital, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Hubei Cancer Hospital, Wuhan
  - Tongji Hospital Tongji Medical College of HUST, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan DY, Liu FR, Wei XL, Luo SX, Zhuang ZX, Wang ZN, Liu FN, Zhang YQ, Yang JW, Chen ZD, Wang YS, Wang JY, Liang XH, Wu XJ, Zheng YL, Liu J, Shi X, Kumar R, Liu W, Chen B, Zhang DS, Xu RH. Claudin 18.2-targeting antibody-drug conjugate CMG901 in patients with advanced gastric or gastro-oesophageal junction cancer (KYM901): a multicentre, open-label, single-arm, phase 1 trial. Lancet Oncol. 2025 Feb;26(2):227-238. doi: 10.1016/S1470-2045(24)00636-3. Epub 2025 Jan 6. PMID 39788133